CLINICAL TRIAL: NCT04313400
Title: A Two Part, Phase I/II, Multi-Center, Double-Blind, Randomized, Vehicle-Controlled Study of the Safety and Efficacy of Topically Applied AMTX-100 CF in Adult Patients With Mild to Moderate Atopic Dermatitis
Brief Title: Topically Applied AMTX-100 CF for Adult Patients With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amytrx Therapeutics, Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMTX100-AD-01
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis
Keywords: AD
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Intervention Model Description: Part 1 (Phase I):
  Part 1 of the study is an open-label, dose-escalation study to determine the MTD of AMTX-100 CF (1.1% w/w) for the highest treated percentage of the BSA affected with AD. Five (5) cohorts will be sequentially enrolled in the Part 1 of the study. Each cohort will include five (5) patients with eligible, treatable percentages of BSA affected with AD.
  Part 2 (Phase II):
  Part 2 of the study is a multi-center, double-blind, randomized, vehicle-controlled, dose-ranging study of the safety and efficacy of topically applied AMTX-100 CF3 in adult patients with Mild to Moderate AD. Sixty (60) patients will be enrolled in 2 groups of AMTX-100 CF3 along with a placebo (vehicle). The patients will be randomized in a 1:1 ratio with thirty (30) subjects in Group A: 1.1% of AMTX-100 CF3 and thirty (30) subjects will be randomized to Group B placebo (vehicle 0% w/w).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 (Phase I) of the study is open-labeled. Part 2 (Phase II) of the study is double-blinded (Masking: Participant, Care Provider, Investigator, and Outcomes Assessor).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Dose Escalation: 3% to 70% of the BSA (Experimental): Open-label, five (5) cohorts were sequentially enrolled. AMTX-100 CF 1.1% w/w, topically applied twice a day for 7 consecutive days to all treatable AD affected areas from 3% to 70% of the Body Surface Area (BSA) (3% BSA ≤ AD Affected Area ≤ 70% BSA)
  Interventions: Drug: 1.1% w/w AMTX-100 CF-part1
- Part 2 Group A: 1.1% w/w (Experimental): AMTX-100 CF3 (1.1% w/w), topically applied twice a day for 28 consecutive days to all treatable AD affected areas
  Interventions: Drug: 1.1% w/w AMTX-100 CF3-part2
- Part 2 Group B: Placebo (Placebo Comparator): Placebo (Vehicle) (0% w/w), topically applied twice a day for 28 consecutive days to all treatable AD affected areas
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 1.1% w/w AMTX-100 CF-part1 — AMTX-100 CF, topical cream with 1.1% w/w active pharmaceutical ingredient
  Arms: Part 1 Dose Escalation: 3% to 70% of the BSA
Drug: Placebo — Topical cream manufactured to mimic AMTX-100 CF3
  Other Names: placebo (vehicle 0% w/w)
  Arms: Part 2 Group B: Placebo
Drug: 1.1% w/w AMTX-100 CF3-part2 — AMTX-100 CF3, topical cream with 1.1% w/w active pharmaceutical ingredient
  Other Names: part2
  Arms: Part 2 Group A: 1.1% w/w

SUMMARY:
This study determines the Maximum Tolerable Dose (MTD) by maximum BSA percentage treated and evaluates safety and efficacy of 1.1% w/w AMTX-100 CF versus placebo (vehicle).

The study has two parts:

Phase I (Part 1):

Approximately Twenty-five (25) subjects with various treatable Body Surface Area (BSA) involvement of Mild to Moderate Atopic Dermatitis will be enrolled in the study and treated with 1.1% w/w AMTX-100 CF.

Phase II (Part 2):

Approximately sixty (60) subjects with Mild to Moderate Atopic Dermatitis with various treatable BSA involvement of Mild to Moderate Atopic Dermatitis will be randomized to be treated with 1.1% w/w AMTX-100 CF3 concentration or Vehicle (Placebo) in the study.

DETAILED DESCRIPTION:
AMTX-100 CF3 drug product is formulated as a water-based, topical cream incorporating a 28-amino acid synthetic polypeptide (AMTX-100) as the active pharmaceutical ingredient (API). AMTX-100 is a chimeric, cell-penetrating, bifunctional nuclear transport modifier (NTM), that is engineered to modulate nuclear transport of transcription factors (NF-κB, NFAT, AP-1, and STAT1) involved in the activation of gene expression of key mediators of inflammation (TNFα, IL-1β, IL-6, IL-17, MCP-1, etc.) and metabolic syndrome (ChREBP and SREBP) by importin α/β complex and importin β, respectively. This further leads to a reduction in pro-inflammatory cytokine/chemokine production and lipid and carbohydrate metabolic products.

AMTX-100 CF3 is intended to improve symptoms associated with mild to moderate Atopic Dermatitis in adults. This Phase I/II study aims to determine the Maximum Tolerable Dose (MTD) by maximum BSA percentage treated and to evaluate efficacy of 1.1% w/w AMTX-100 CF3 versus placebo (vehicle).

ELIGIBILITY:
Part 1 Inclusion Criteria:

Subjects are required to meet ALL of the following criteria for enrollment into the Phase I (Part 1) of the study:

1. Male or female subjects who are 18 years or older
2. If female and not infertile (defined below), the subject must agree for the duration of the study to use one of the following forms of contraception 1) systemic hormonal treatment 2) an intrauterine device (IUD) which was implanted at least 2 months prior to screening or 3) "double-barrier" contraception (condom, diaphragm and spermicide are each considered a barrier). Females are considered to be infertile if they are either a) surgically sterile or b) have had spontaneous amenorrhea for at least the last 2 years and at least 2 years after the onset of amenorrhea while not receiving hormone replacement therapy and had a Follicle-Stimulating Hormone (FSH) level greater than 40 mIU/mL and an estradiol level less than 30 pg/mL
3. All fertile female subjects as described above need to have a negative urine pregnancy test at the screening and baseline visits
4. Subject is capable of providing informed consent and is willing to sign the ICF prior to study Screening and agrees to comply with the study protocol requirements
5. Subject is able to apply topical products on all treatable assigned areas by self and/or caregiver (if applicable), per the Investigator
6. Subject is in general good physical/mental health per the Investigator
7. Subject's Total Body Surface Area (BSA) is between 1.5 and 2.1 m2 per the Mosteller formula
8. The subject has physician confirmed mild to moderate Atopic Dermatitis (AD) defined by the Eichenfield revised criteria of Hannifin and Rajka, for at least 6 months prior to study enrollment
9. Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD™) score of 2 or 3 (mild to moderate) at the screening and baseline visits
10. Subject has Atopic Dermatitis (AD) involvement with eligible treatable percent of the BSA appropriate for topical treatment per the assigned cohort at the screening and baseline visits per below:

    1. Cohort 1: 3% BSA ≤ AD Affected Area ≤ 6% BSA
    2. Cohort 2: 6% BSA < AD Affected Area ≤ 12% BSA
    3. Cohort 3: 12% BSA < AD Affected Area ≤ 24% BSA
    4. Cohort 4: 24% BSA < AD Affected Area ≤ 48% BSA
    5. Cohort 5: 48% BSA < AD Affected Area ≤ 70% BSA

Note: Calculation of Treatable BSA percentage (% of the total BSA that is AD-involved, excluding the scalp, face, eyes, eyelids, neck, hands, palms, feet, groin, genitals or axillae) will be completed by the method below:

o "Handprint Method": the area represented by the palm with all five digits adducted together is approximately 1% of the subject's BSA

Part 1 Exclusion Criteria:

Subjects are required to meet NONE of the following criteria for enrollment into the Phase I (Part 1) of the study:

1. Pregnant or lactating females or women who are planning for pregnancy in the next 6 months
2. Women at postpartum for 3 months or less prior to screening
3. Serious medical illnesses such as end-stage renal disease, liver failure or heart failure that, in the opinion of the Investigator may interfere with the conduct of the study
4. Subjects with abnormal vital signs, physical and dermatological exams or clinical laboratory evaluations considered clinically significant by the Principal Investigator, which in the opinion of the PI would significantly interfere with the study conduct
5. Subjects with any concurrent skin condition that could interfere with the evaluation of the treatment areas, as determined by the investigator
6. The subject has a planned major surgical intervention for a pre-existing condition within the duration of the study
7. The subject has a history of drug or alcohol abuse that would impair or risk the subject's full participation in the study, in the opinion of the investigator.
8. Participation in a clinical trial within 3 months, or more than two clinical trials within 12 months prior to screening
9. Concurrent or recent use of topical steroids, topical immunosuppressive/immunomodulative drugs, topical vitamin D3 derivative, topical retinoids, anthralin, coal tar (except when used as shampoo) or salicylic acid within 14 days of the baseline visit
10. The subject has severe AD as determined by vIGA-AD™ score higher than 3
11. The subject cannot avoid systemic treatments (including systemic corticosteroids, immunotherapy, biologics or phototherapy) for AD during the study per the Investigator
12. The subject has previously received any systemic treatments, immunotherapy, biologics or phototherapy for AD within 12 months prior to study enrollment
13. Current or expected use of prohibited medications as described in Section 7, unless approved by the study Medical Monitor
14. The subject has concurrent contact dermatitis or history of anaphylactic reaction

Part 2 Inclusion Criteria:

Subjects are required to meet ALL of the following criteria for randomization into the Phase II (Part 2) of the study:

1. Male or female subjects who are 18 years or older.
2. If female and not infertile (defined below), the subject must agree for the duration of the study to use one of the following forms of contraception 1) systemic hormonal treatment 2) an intrauterine device (IUD) which was implanted at least 2 months prior to screening or 3) "double-barrier" contraception (condom, diaphragm and spermicide are each considered a barrier). Females are considered to be infertile if they are either a) surgically sterile or b) have had spontaneous amenorrhea for at least the last 2 years and at least 2 years after the onset of amenorrhea while not receiving hormone replacement therapy.
3. All fertile female subjects as described above need to have a negative urine pregnancy test at the screening and baseline visits.
4. Subject is capable of providing informed consent and is willing to sign the ICF prior to study Screening and agrees to comply with the study protocol requirements.
5. Subject is able to apply topical products on all the treatable areas by self and/or caregiver (if applicable), per the Investigator.
6. Subject is willing and able to comply with all clinic visits and study-related procedures.
7. Subject is able to understand and complete study-related questionnaires.
8. The subject has physician confirmed mild to moderate Atopic Dermatitis (AD) defined by the Eichenfield revised criteria of Hannifin and Rajka, for at least 6 months prior to study enrollment.
9. Validated Investigator's Global Assessment for Atopic Dermatitis (vIGA-AD™) score of 2 or 3 (mild to moderate) at the screening and baseline visits.
10. Eczema Area and Severity Index (EASI) score lower than 23 at the screening and baseline visits
11. Subject has Atopic Dermatitis (AD) involvement of between 5% and 30% of the treatable BSA (excluding the scalp, face, eyes, eyelids, hands, palms, feet, groin, genitals or the axillae) appropriate for topical treatment at the screening and baseline visits.

    Note: Calculation of Treatable BSA percentage (% of the total BSA that is AD-involved, excluding the scalp, face, eyes, eyelids, hands, palms, feet, groin, genitals or the axillae) will be completed by the "Rule of Nines" method:

    o Where values of 9% or 18% of BSA are assigned to specific regions in the adult subject (head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%])
12. Subjects must be applying stable doses of an additive-free, basic bland emollient twice-daily for at least 1 week immediately before the baseline visit (Visit 2, Day 0), and to be continued throughout the study.

Note: The additive-free, basic bland emollients should be applied no earlier than 1 hour before or after the administration of the study treatment.

Part 2 Exclusion Criteria:

Subjects are required to meet NONE of the following criteria for randomization into the Phase II (Part 2) of the study:

1. Pregnant or lactating females or women who are planning for pregnancy in the next 6 months
2. Women at postpartum for 3 months or less prior to screening
3. Serious medical illnesses such as end-stage renal disease, liver failure or heart failure that, in the opinion of the Investigator may interfere with the conduct of the study
4. Subjects with abnormal vital signs, physical and dermatological exams or clinical laboratory evaluations considered clinically significant by the Principal Investigator, which in the opinion of the PI would significantly interfere with the study conduct
5. Subjects with any concurrent skin condition that could interfere with the evaluation of the treatment areas, as determined by the investigator
6. The subject has a planned major surgical intervention for a pre-existing condition within the duration of the study
7. The subject has a history of drug or alcohol abuse that would impair or risk the subject's full participation in the study, in the opinion of the investigator.
8. Participation in a clinical trial within 3 months, or more than two clinical trials within 12 months prior to screening
9. Concurrent or recent use of prescription moisturizers, topical steroids, topical immunosuppressive/immunomodulative drugs, topical vitamin D3 derivative, topical retinoids, anthralin, coal tar (except when used as shampoo) or salicylic acid within 14 days of the baseline visit
10. The subject has severe AD as determined by vIGA-AD™ score higher than 3
11. The subject cannot avoid systemic treatments (including systemic corticosteroids, immunotherapy, biologics or phototherapy) for AD during the study per the Investigator
12. The subject has previously received any systemic treatments, immunotherapy, biologics or phototherapy for AD within 12 months prior to study enrollment
13. Current or expected use of prohibited medications and procedures during study treatment, as described in Section 7, unless approved by the study Medical Monitor
14. Subject has unstable AD or any consistent requirement for high-potency topical corticosteroids to manage AD signs and symptoms
15. Subject has a significant active systemic or localized infection, including known actively infected AD
16. Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks of the screening visit
17. The subject has previously received AMTX-100 CF
18. Subject has any other medical or psychological condition (including relevant laboratory abnormalities at screening) that, in the opinion of the investigator, may suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the study patient as a result of his/her participation in this clinical trial, may make patient's participation unreliable, or may interfere with study assessments
19. The subject has concurrent contact dermatitis; or history of anaphylactic reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arezou Bayat, MD, MPH, Study Director — Amarex Clinical Research, LLC (Amarex)
Locations (11):
- United States (11):
  - Amytrx Investigational site, Cerritos, California
  - Amytrx Investigational site, Encino, California
  - Amytrx Investigational site, Long Beach, California
  - Amytrx Investigational site, North Hollywood, California
  - Amytrx Investigational site, San Diego, California
  - Amytrx Investigational site, Sherman Oaks, California
  - Amytrx Investigational site, Miami, Florida
  - Amytrx Investigational site, Miramar, Florida
  - Amytrx Investigational site, Troy, Michigan
  - Amytrx Investigational site, New York, New York
  - Amytrx Investigational site, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Qiao H, Zienkiewicz J, Hawiger J. Anti-inflammatory control of human skin keratinocytes by targeting nuclear transport checkpoint. Skin Health Dis. 2024 Mar 3;4(3):e356. doi: 10.1002/ski2.356. eCollection 2024 Jun. PMID 38846687
- [Derived] Liu Y, Zienkiewicz J, Qiao H, Gibson-Corley KN, Boyd KL, Veach RA, Hawiger J. Genomic control of inflammation in experimental atopic dermatitis. Sci Rep. 2022 Nov 7;12(1):18891. doi: 10.1038/s41598-022-23042-x. PMID 36344555

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 Dose Escalation: Cohort 1: Open-label AMTX-100 CF 1.1% w/w, topically applied twice a day for seven consecutive days to all treatable AD affected areas of 3-6% of the BSA (3% BSA ≤ AD Affected Area ≤ 6% BSA)
- Part 1 Dose Escalation: Cohort 2: Open-label AMTX-100 CF 1.1% w/w, topically applied twice a day for seven consecutive days to all treatable AD affected areas of 6-12% of the BSA (6% BSA < AD Affected Area ≤ 12% BSA)
- Part 1 Dose Escalation: Cohort 3: Open-label AMTX-100 CF 1.1% w/w, topically applied twice a day for seven consecutive days to all treatable AD affected areas of 12-24% of the BSA (12% BSA < AD Affected Area ≤ 24% BSA)
- Part 1 Dose Escalation: Cohort 4: Open-label AMTX-100 CF 1.1% w/w, topically applied twice a day for seven consecutive days to all treatable AD affected areas of 24-48% of the BSA (24% BSA < AD Affected Area ≤ 48% BSA)
- Part 1 Dose Escalation: Cohort 5: Open-label AMTX-100 CF 1.1% w/w, topically applied twice a day for seven consecutive days to all treatable AD affected areas of 48-70% of the BSA (48% BSA < AD Affected Area ≤ 70% BSA)
Period: Overall Study
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 1 Dose Escalation: Cohort 4 | Part 1 Dose Escalation: Cohort 5 | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Started | 5 | 5 | 5 | 4 | 7 | 33 | 32
Completed (These data refer only to completing treatment.) | 5 | 5 | 5 | 4 | 7 | 27 | 31
Not Completed | 0 | 0 | 0 | 0 | 0 | 6 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 4 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 1 Dose Escalation: Cohort 4 | Part 1 Dose Escalation: Cohort 5 | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 7 | 33 | 32 | 91
Age, Continuous [Mean (Full Range); unit: years] | 51.6 [24.0 to 74.0] | 41.4 [20.0 to 59.0] | 40.6 [20.0 to 57.0] | 62.8 [40.0 to 74.0] | 49.4 [22.0 to 75.0] | 46.1 [18.0 to 74.0] | 46.0 [18.0 to 90.0] | 47.35 [18.0 to 90.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 1 | 4 | 20 | 17 | 49
  Male | 1 | 4 | 3 | 3 | 3 | 13 | 15 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 0 | 10 | 13 | 27
  Not Hispanic or Latino | 4 | 4 | 4 | 3 | 7 | 23 | 19 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 7 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 2 | 2 | 5 | 10 | 5 | 30
  White | 3 | 1 | 3 | 2 | 1 | 13 | 20 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 5
Height (cm) [Mean (Full Range); unit: centimeter] | 162.7 [153.5 to 175.0] | 171.9 [165.0 to 182.5] | 168.0 [155.0 to 182.5] | 169.3 [155.0 to 179.1] | 167.7 [157.4 to 182.0] | 167.5 [143.0 to 190.5] | 168.6 [155.0 to 188.0] | 167.95 [143.0 to 190.5]
Weight (kg) [Mean (Full Range); unit: Kilogram] | 69.0 [63.0 to 79.0] | 88.9 [65.0 to 120.5] | 64.5 [46.5 to 86.0] | 75.4 [60.3 to 90.8] | 80.2 [56.5 to 103.0] | 81.2 [46.2 to 134.1] | 82.3 [54.4 to 121.3] | 78.85 [46.2 to 134.1]
BMI (kg/m2) [Mean (Full Range); unit: kilogram per meter squared] | 26.1 [22.0 to 30.9] | 30.1 [21.5 to 40.7] | 23.1 [15.3 to 32.6] | 26.2 [23.2 to 30.3] | 28.6 [20.7 to 34.6] | 28.9 [17.8 to 52.4] | 28.9 [20.0 to 42.2] | 27.95 [15.3 to 52.4]
BSA (m2) [Mean (Full Range); unit: meter squared] | 1.8 [1.6 to 1.9] | 2.0 [1.7 to 2.4] | 1.7 [1.4 to 2.0] | 1.9 [1.6 to 2.1] | 1.9 [1.6 to 2.2] | 1.9 [1.4 to 2.4] | 2.0 [1.6 to 2.4] | 1.9 [1.4 to 2.4]

OUTCOME MEASURES:

1. Primary Outcome: Part 1 (Phase I) Primary: Maximum Tolerable Dose
Description: Maximum Tolerable Dose (MTD) by maximum percentage of Body Surface Area (BSA) treated, by evaluation of dose-limiting toxicity (DLT) of AMTX-100 CF (1.1% w/w concentration) based on the safety profile
Time Frame: Over the 7-day treatment period
Measure: Number; unit: Grams of IP per application
Arm/Group | Part 1 Dose Escalation: 3% to 70% of the BSA
Number analyzed (Participants) | 26
Grams of IP per application | 29.2

2. Primary Outcome: Part 2 (Phase II) Primary: Proportion of Responder Subjects at Day 28
Description: Proportion of responder subjects at Day 28, defined as subjects with both Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD™) score of 0 (clear) or 1 (almost clear) (on a 5-point scale) and a reduction of ≥ 2 points from baseline
  Note: Subjects who have received rescue treatments will be considered non-responders
  Note: We acknowledge that the "percentage" was reported, while the outcome measure indicates "proportion". It was concluded that using "percentage" represents the results more apparent.
Time Frame: Day 28
Population: There were missing subjects in both groups.
Measure: Number; unit: Percentage of Responder Subjects
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 26 | 31
Percentage of Responder Subjects | 3.8 | 9.7

3. Secondary Outcome: Part 2 (Phase II) Secondary Efficacy Endpoints: Percent Change From Baseline in vIGA-AD™ at Days 7, 14, 21, 28, and 42
Description: The 5-point Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD™) is a validated measure of disease severity and success of atopic dermatitis treatments in clinical trials. The ratings (0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe) are an overall assessment of AD skin lesions, based on the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Baseline to Days 7, 14, 21, 28, and 42
Population: There were missing subjects in both groups.
Measure: Mean (Standard Deviation); unit: percentage of vIGA-AD change at visits
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 33 | 32
percentage of vIGA-AD change at visits
  Visit 3 (Day 7): number analyzed (Participants) | 32 | 32
  Visit 3 (Day 7) | -2.6 (14.73) | -5.7 (13.79)
  Visit 4 (Day 14): number analyzed (Participants) | 30 | 32
  Visit 4 (Day 14) | -6.1 (16.66) | -11.5 (19.6)
  Visit 5 (Day 21): number analyzed (Participants) | 28 | 32
  Visit 5 (Day 21) | -11.9 (22.16) | -14.1 (22.44)
  End of Treatment (Day 28): number analyzed (Participants) | 26 | 31
  End of Treatment (Day 28) | -14.1 (26.54) | -20.4 (27.79)
  Follow-Up (Day 42): number analyzed (Participants) | 27 | 30
  Follow-Up (Day 42) | -16.7 (30.31) | -26.1 (34.93)

4. Secondary Outcome: Part 2 (Phase II) Secondary Efficacy Endpoints: Proportion of Subjects at Days 7, 14, 21, 28, and 42 With Both vIGA-AD™ Score of 0 (Clear) or 1 (Almost Clear) on a 5-point Scale and a Reduction of ≥ 1 Point From Baseline
Description: The 5-point Validated Investigator Global Assessment scale for Atopic Dermatitis (vIGA-AD™) is a validated measure of disease severity and success of atopic dermatitis treatments in clinical trials. The ratings (0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe) are an overall assessment of AD skin lesions, based on the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
  Note: We acknowledge that the "percentage" is reported, while the outcome measure indicates "proportion". It was concluded that using "percentage" represents the results more apparent.
Time Frame: Days 7, 14, 21, and 28
Population: There were missing subjects in both groups.
Measure: Number; unit: Percent of Subjects With vIGA-AD of 0/1
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 33 | 32
Percent of Subjects With vIGA-AD of 0/1
  Visit 3 (Day 7): number analyzed (Participants) | 32 | 32
  Visit 3 (Day 7) | 0 | 3.1
  Visit 4 (Day 14): number analyzed (Participants) | 30 | 32
  Visit 4 (Day 14) | 6.7 | 9.4
  Visit 5 (Day 21): number analyzed (Participants) | 28 | 32
  Visit 5 (Day 21) | 14.3 | 12.5
  End of Treatment (Day 28): number analyzed (Participants) | 26 | 31
  End of Treatment (Day 28) | 11.5 | 25.8

5. Secondary Outcome: Part 2 (Phase II) Secondary Efficacy Endpoints: Percent Change From Baseline in Eczema Area and Severity Index (EASI) at Days 7, 14, 21, 28 and 42
Description: The Eczema Area and Severity Index (EASI) is a validated measure to assess the severity and extent of AD (Hanifin et al., 2001). The EASI is a composite index with scores ranging from 0 to 72, where a higher score indicates increased extent and severity of atopic dermatitis.
Time Frame: Baseline to Days 7, 14, 21, 28, and 42
Population: There were missing subjects in both groups.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline in EASI
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 33 | 32
Percent Change from Baseline in EASI
  Visit 3 (Day 7): number analyzed (Participants) | 32 | 32
  Visit 3 (Day 7) | -7.7 (21.4) | -10.7 (19.13)
  Visit 4 (Day 14): number analyzed (Participants) | 30 | 32
  Visit 4 (Day 14) | -16.0 (22.55) | -20.9 (29.27)
  Visit 5 (Day 21): number analyzed (Participants) | 28 | 32
  Visit 5 (Day 21) | -29.0 (28.7) | -23.7 (35.17)
  End of Treatment (Day 28): number analyzed (Participants) | 26 | 31
  End of Treatment (Day 28) | -29.9 (32.98) | -34.5 (43.29)
  Follow-Up (Day 42): number analyzed (Participants) | 27 | 30
  Follow-Up (Day 42) | -32.5 (39.02) | -41.9 (38.27)

6. Secondary Outcome: Part 2 (Phase II) Secondary Efficacy Endpoints: Proportion of Subjects With EASI-75, Defined as Achieving at Least a 75% Reduction From Baseline in EASI at Days 7, 14, 21, 28, and 42
Description: The Eczema Area and Severity Index (EASI) is a validated measure to assess the severity and extent of AD. The EASI is a composite index with scores ranging from 0 to 72, where a higher score indicates increased extent and severity of atopic dermatitis.
  Note: We acknowledge that the "percentage" is reported, while the outcome measure indicates "proportion". It was concluded that using "percentage" represents the results more apparent.
Time Frame: Days 7, 14, 21, 28, and 42
Population: There were missing subjects in both groups.
Measure: Number; unit: Percentage of Subjects With EASI-75
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 33 | 32
Percentage of Subjects With EASI-75
  Visit 3 (Day 7): number analyzed (Participants) | 32 | 32
  Visit 3 (Day 7) | 3.1 | 3.1
  Visit 4 (Day 14): number analyzed (Participants) | 30 | 32
  Visit 4 (Day 14) | 3.3 | 3.1
  Visit 5 (Day 21): number analyzed (Participants) | 28 | 32
  Visit 5 (Day 21) | 7.1 | 9.4
  End of Treatment (Day 28): number analyzed (Participants) | 26 | 31
  End of Treatment (Day 28) | 7.7 | 12.9
  Follow-Up (Day 42): number analyzed (Participants) | 27 | 30
  Follow-Up (Day 42) | 14.8 | 20.0

7. Secondary Outcome: Part 2 (Phase II) Secondary Efficacy Endpoints: Proportion of Subjects With EASI-50, Defined as Achieving at Least a 50% Reduction From Baseline in EASI at Days 7, 14, 21, 28, and 42
Description: as for outcome 6
Time Frame: Days 7, 14, 21, 28, and 42
Population: There were missing subjects in both groups.
Measure: Number; unit: Percentage of Subjects With EASI-50
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 33 | 32
Percentage of Subjects With EASI-50
  Visit 3 (Day 7): number analyzed (Participants) | 32 | 32
  Visit 3 (Day 7) | 6.3 | 3.1
  Visit 4 (Day 14): number analyzed (Participants) | 30 | 32
  Visit 4 (Day 14) | 10.0 | 21.9
  Visit 5 (Day 21): number analyzed (Participants) | 28 | 32
  Visit 5 (Day 21) | 25.0 | 28.1
  End of Treatment (Day 28): number analyzed (Participants) | 26 | 31
  End of Treatment (Day 28) | 26.9 | 45.2
  Follow-Up (Day 42): number analyzed (Participants) | 27 | 30
  Follow-Up (Day 42) | 25.9 | 46.7

8. Secondary Outcome: Part 2 (Phase II) Secondary Efficacy Endpoints: Percent Change From Baseline in Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) at Days 7, 14, 21, 28, and 42
Description: The Pruritus Numeric Rating Scale (NRS) is a simple assessment tool that subjects used to report the intensity of their pruritus (itch) during a daily recall period. Subjects were asked the following questions:
  • For maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?"
  Note: The weekly average of peak daily pruritus NRS was calculated by summing the daily scores for a week and dividing by the number of days with recorded scores, resulting in a range of 0 to 10.
Time Frame: Baseline, Days 7, 14, 21, 28 and 42
Population: There were missing subjects in both groups.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline in NRS
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 33 | 32
Percent Change from Baseline in NRS
  Visit 3 (Day 7): number analyzed (Participants) | 32 | 31
  Visit 3 (Day 7) | -15.1 (28.15) | -9.9 (17.22)
  Visit 4 (Day 14): number analyzed (Participants) | 29 | 30
  Visit 4 (Day 14) | -17.1 (40.83) | -8.5 (37.26)
  Visit 5 (Day 21): number analyzed (Participants) | 27 | 31
  Visit 5 (Day 21) | -22.8 (43.81) | -18.7 (26.88)
  End of Treatment (Day 28): number analyzed (Participants) | 27 | 30
  End of Treatment (Day 28) | -25.8 (47.12) | -25.2 (36.25)
  Follow-Up (Day 42): number analyzed (Participants) | 25 | 28
  Follow-Up (Day 42) | -27.6 (45.28) | -38.4 (27.24)

9. Secondary Outcome: Part 2 (Phase II) Secondary Efficacy Endpoints: Proportion of Subjects With Improvement (Reduction) of Weekly Average of Peak Daily Pruritus NRS ≥ 3 From Baseline at Day 28 and 42
Description: The Pruritus Numeric Rating Scale (NRS) is a simple assessment tool that subjects used to report the intensity of their pruritus (itch) during a daily recall period. Subjects were asked the following questions:
  • For maximum itch intensity: "On a scale of 0 to 10, with 0 being 'no itch' and 10 being the 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?"
  Note: The weekly average of peak daily pruritus NRS was calculated by summing the daily scores for a week and dividing by the number of days with recorded scores, resulting in a range of 0 to 10.
  Note: We acknowledge that the "percentage" is reported, while the outcome measure indicates "proportion". It was concluded that using "percentage" represents the results more apparent.
Time Frame: Days 28 and 42
Population: There were missing subjects in both groups.
Measure: Number; unit: Percentage of Subjects with Improved NRS
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 33 | 32
Percentage of Subjects with Improved NRS
  End of Treatment (Day 28): number analyzed (Participants) | 27 | 31
  End of Treatment (Day 28) | 18.5 | 32.3
  Follow-Up (Day 42): number analyzed (Participants) | 25 | 29
  Follow-Up (Day 42) | 20.0 | 34.5

10. Secondary Outcome: Part 2 (Phase II) Secondary Efficacy Endpoints: Percent Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Day 28
Description: The Dermatology Life Quality Index (DLQI) is a 10-item, validated questionnaire to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The format is a simple response (0 to 3 where 0 is "not at all" and 3 is "very much") to 10 questions, which assess QOL over the past week, with an overall scoring system of 0 to 30. A high score is indicative of a poor QOL. For general inflammatory skin conditions, a change in DLQI score of at least 4 points is considered clinically important
Time Frame: Baseline, Day 28
Population: There were missing subjects in both groups.
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline in DLQI
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 24 | 30
Percent Change from Baseline in DLQI | -26.6 (42.14) | -36.3 (75.35)

11. Secondary Outcome: Part 2 (Phase II) Secondary Efficacy Endpoints: Percent Change From Baseline of the Treated BSA With Active AD at Day 28, and 42
Description: For Part 2, BSA affected by AD was assessed by the investigator per calculation of treatable % BSA by the "Rule of Nines" method:
  Values of 9% or 18% of surface area are assigned to specific regions in the adult (head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%])
Time Frame: Baseline, Days 28, and 42
Population: There were missing subjects in both groups.
Measure: Mean (Standard Deviation); unit: Percent Change of the Treated BSA
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 33 | 32
Percent Change of the Treated BSA
  End of Treatment (Day 28): number analyzed (Participants) | 26 | 31
  End of Treatment (Day 28) | -27.6 (35.72) | -26.9 (33.16)
  Follow-Up (Day 42): number analyzed (Participants) | 27 | 30
  Follow-Up (Day 42) | -32.8 (36.03) | -33.7 (36.04)

12. Other Pre Specified Outcome: Part 1 (Phase I) Exploratory Outcome Measures: Percent Change From Baseline of the Treated BSA With Active AD at Day 7
Description: For Part 1, Body surface area (BSA) affected by AD was assessed by the investigator per calculation of treatable % BSA by the handprint method:
  "Handprint Method": the area represented by the palm with all five digits adducted together is approximately 1% of the subject's BSA
Time Frame: Baseline, Day 7
Measure: Mean (Standard Deviation); unit: percent change at the End of Treatment
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 1 Dose Escalation: Cohort 4 | Part 1 Dose Escalation: Cohort 5
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 7
percent change at the End of Treatment | -46.7 (30.91) | -44.3 (44.15) | -43.3 (44.62) | -38.1 (28.84) | -21.7 (32.31)

13. Other Pre Specified Outcome: Part 1 (Phase I) Exploratory Outcome Measures: Change From Baseline in Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD™) at Day 7
Description: as for outcome 3
Time Frame: Baseline, Day 7
Measure: Number; unit: number of subjects
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 1 Dose Escalation: Cohort 4 | Part 1 Dose Escalation: Cohort 5
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 7
number of subjects
  Baseline-Mild | 5 | 4 | 1 | 1 | 0
  Baseline-Moderate | 0 | 1 | 4 | 3 | 7
  End of Treatment-Clear | 1 | 1 | 1 | 0 | 0
  End of Treatment-Almost Clear | 3 | 3 | 2 | 1 | 1
  End of Treatment-Mild | 1 | 0 | 0 | 2 | 2
  End of Treatment-Moderate | 0 | 1 | 2 | 1 | 4

14. Other Pre Specified Outcome: Part 1 (Phase I) Safety Outcome Measures: Incidence of Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavorable or unintended sign, symptom, or disease that occurred or was reported by the subject to have occurred, or a worsening of a pre-existing condition. Treatment Emergent Adverse Events (TEAEs) were defined as adverse events with onset date on or after the first treatment.
Time Frame: Baseline through follow-up (Day 21)
Measure: Number; unit: number of events
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 1 Dose Escalation: Cohort 4 | Part 1 Dose Escalation: Cohort 5
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 7
number of events
  Any TEAE | 1 | 3 | 3 | 0 | 2
  Any Related TEAE | 0 | 0 | 0 | 0 | 0

15. Other Pre Specified Outcome: Part 2 (Phase II) Safety Outcome Measures: Incidence of Treatment-Emergent Adverse Events (TEAEs)
Description: as for outcome 14
Time Frame: Baseline through follow-up (Day 42)
Measure: Number; unit: number of events
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 33 | 32
number of events
  Any TEAE | 12 | 3
  Any Related TEAE | 2 | 1

16. Other Pre Specified Outcome: Part 2 (Phase II) Safety Outcome Measures: Incidence of Withdrawals From the Study Due to TEAEs
Description: as for outcome 14
Time Frame: Baseline through follow-up (Day 42)
Measure: Number; unit: number of subjects
Arm/Group | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
Number analyzed (Participants) | 33 | 32
number of subjects | 1 | 1

17. Other Pre Specified Outcome: Part 1 (Phase I) Safety Outcome Measures: Incidence of Withdrawals From the Study Due to TEAEs
Description: as for outcome 14
Time Frame: Baseline through follow-up (Day 21)
Measure: Number; unit: number of subjects
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 1 Dose Escalation: Cohort 4 | Part 1 Dose Escalation: Cohort 5
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 7
number of subjects | 0 | 0 | 0 | 0 | 0

18. Other Pre Specified Outcome: Part 1 (Phase I) Safety Outcome Measures: Changes in Study Treatment Application Site Reaction Assessment
Description: Tolerability of topically applied AMTX-100 CF was evaluated based on investigator-assessed application site reactions assessment. Local skin reactions were assessed in all areas treated with AMTX-100 CF and graded by the investigator on a scale of 0 to 4 based on the area with the most severe skin reaction among all treated areas. A grade of 0 represented no reaction, and a grade of 4 indicated a marked and severe skin reaction that extended beyond the treated areas.
Time Frame: Baseline (post-dose), End of Treatment (Day 7), and Follow-up (Day 21)
Measure: Mean (Standard Deviation); unit: Units on an ordinal scale
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 1 Dose Escalation: Cohort 4 | Part 1 Dose Escalation: Cohort 5
Number analyzed (Participants) | 5 | 5 | 5 | 4 | 7
Units on an ordinal scale
  Baseline (Post-dose) | -0.2 (1.64) | -0.4 (1.14) | -1.8 (0.84) | -2.0 (2.16) | -0.9 (0.9)
  End of Treatment (Day 7) | -0.8 (1.64) | -0.6 (1.52) | -3.0 (3.16) | -4.8 (5.91) | -1.4 (1.40)
  Follow-Up (Day 21) | -1.0 (1.73) | -1.8 (2.77) | -4.4 (3.91) | -4.5 (3.51) | -1.6 (2.37)

ADVERSE EVENTS:
Time Frame: Phase I (Part 1) Baseline through follow-up (Day 21) Phase II (Part 2) Baseline through follow-up (Day 42)
Description: An adverse event (AE) may or may not be related to the study treatment. All AEs were elicited through direct questioning and subject reports. Any abnormality in physical examination findings or laboratory results that the investigator believes is clinically significant (CS) to the research subject and that occurred after initiation of the first study treatment was reported as AEs. Abnormal findings that were not CS were not recorded as an AE.
Arm/Group | Part 1 Dose Escalation: Cohort 1 | Part 1 Dose Escalation: Cohort 2 | Part 1 Dose Escalation: Cohort 3 | Part 1 Dose Escalation: Cohort 4 | Part 1 Dose Escalation: Cohort 5 | Part 2 Group A: 1.1% w/w | Part 2 Group B: Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/4 | 0/7 | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/4 | 0/7 | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 1/5 | 3/5 | 2/5 | 0/4 | 2/7 | 5/33 | 3/32
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Dose Escalation: Cohort 1 (N=5) | Part 1 Dose Escalation: Cohort 2 (N=5) | Part 1 Dose Escalation: Cohort 3 (N=5) | Part 1 Dose Escalation: Cohort 4 (N=4) | Part 1 Dose Escalation: Cohort 5 (N=7) | Part 2 Group A: 1.1% w/w (N=33) | Part 2 Group B: Placebo (N=32)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application Site Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application Site Pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — for the case of this study the term "Dermatitis Atopic" refers to "worsening atopic dermatitis"
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator will refer to the Investigator agreement and clinical trial agreement for the publication and disclosure policy.

DOCUMENTS (5):
  • Study Protocol (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT04313400/Prot_000.pdf
  • Statistical Analysis Plan: Part 2 (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/00/NCT04313400/SAP_001.pdf
  • Statistical Analysis Plan: Part 1 (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT04313400/SAP_002.pdf
  • Informed Consent Form: Part 1 (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT04313400/ICF_003.pdf
  • Informed Consent Form: Part 2 (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT04313400/ICF_004.pdf